CLINICAL TRIAL: NCT06162390
Title: Optimal Concentration of Remifentanil for Achieving Excellent Intubating Condition During Low-dose Neuromuscular Blocking Agent Administration for Intraoperative Neuromonitoring Using Nerve Integrity Monitoring Tube
Brief Title: Optimal Concentration of Remifentanil for NIM Tube Intubation With Low-dose NMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Responsible Party: Principal Investigator, Sung Hye Byun, Associate Professor, Kyungpook National University Chilgok Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: KNUCH 2023-10-033
Record Dates: First submitted 2023-11-20; First posted 2023-12-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Thyroidectomy
Keywords: Intraoperative nerve monitoring; Neuromuscular blocking agents; Remifentanil
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Masking Description: This is one arm non-randomized approach. Since it is a sequential approach of medication administration, the anesthesiologist and patients were blinded to whatever dose was given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remifentanil for NIM tube intubation (Experimental)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Following a sequential allocation scheme, the predetermined Ce of remifentanil for each patient will be determined by the Dixon up-and-down method. The Ce of remifentanil for the first patient will be 4.0 ng/ml, and then the remifentanil Ce will be increased or decreased in 0.5 ng/ml increments for subsequent patients depending on the success or failure of intubation.
  The Ce of remifentanil to provide acceptable intubation at low dose neuromuscular blockade, the primary outcome, will be determined by obtaining seven crossovers of patients with "acceptable intubation"/"unacceptable intubation" and then calculating the mean of the midpoint doses for each independent pair of patients. According to previous studies that estimated EC50 by Dixon's up-and-down method, 6-8 "failure/success crossover pairs" are required, so this study aims to collect independent data of 7 pairs of "intubation acceptable/unacceptable" patients.

SUMMARY:
During thyroid surgery, Intraoperative Neuromonitoring (IONM) plays a crucial role in preventing serious complications such as bilateral vocal cord paralysis. It achieves this by detecting damage to the recurrent laryngeal nerve (RLN) and predicting the RLN's functional status. The utilization of Nerve Integrity Monitoring tubes (NIM tubes) is on the rise for effective IONM. As IONM relies on observing electromyographic (EMG) responses to direct electrical nerve stimulation, the routine use of neuromuscular blocking agents (NMBAs) in general anesthesia can impact the interpretation of IONM results and potentially reduce sensitivity to nerve responses to stimulation. However, the use of NMBAs is essential for ensuring smooth endotracheal intubation in patients undergoing general anesthesia. Numerous studies suggest that NMBA usage provides superior intubation conditions and reduces vocal cord complications compared to scenarios without NMBA.

Various regimens for neuromuscular blockade methods are employed during IONM in thyroid surgery, ranging from not using NMBAs at all to using a full dose of NMBA for intubation. This is followed by the administration of sugammadex, an NMBA reversal agent, before nerve monitoring. One of the methods known for providing satisfactory intubation conditions while ensuring the quality of EMG signals during IONM in thyroid surgery is using rocuronium at an ED95 dose of 0.3 mg/kg. This approach is considered suitable for most IONM scenarios. However, when adequate muscle relaxation is not achieved, not all patients can undergo intubation, necessitating a strategy for appropriate intubation conditions.

Historically, it has been reported that achieving satisfactory intubation conditions without the use of NMBA during general anesthesia requires higher amounts of propofol and opioids. Therefore, the assumption is made that using remifentanil, an opioid used in total intravenous anesthesia (TIVA), at an appropriate concentration can provide acceptable intubation conditions with minimal NMBA use for patients undergoing IONM.

This study aims to determine the optimal concentration of remifentanil needed to achieve excellent intubation conditions in patients undergoing thyroid surgery with IONM using rocuronium 0.3 mg/kg as the NMBA during TIVA

ELIGIBILITY:
Inclusion Criteria:

* All female aged 20-60
* ASA (American Society of Anesthesiologists) physical status I or II
* who scheduled for thyroidectomy under intraoperative neuromonitoring with a nerve integrity monitoring tube (NIM tube)

Exclusion Criteria:

* Patients anticipated to experience challenging intubation.
* Patients who have had an upper respiratory tract infection within the past 2 weeks.
* Patients with a history of heart, lung, and kidney diseases.
* Patients with a body mass index (BMI) of 30 kg/m² or higher.
* Patients currently taking analgesics.
* Patients expressing a desire not to participate in the study.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Optimal effect-site concentration (Ce) of remifentanil | During the tracheal intubation
  Finding the Ce of remifentanil that provides acceptable condition of tracheal intubation when administering a low-dose NMBA is the aim of the study. The Ce of remifentanil for the first patient is 4.0 ng/ml, and then the Ce is increased or decreased in 0.5 ng/ml increments for subsequent patients depending on the success or failure of intubation. About 3 minutes after administering rocuronium 0.3 mg/kg, NIM tube will be intubated. At this time, the intubation condition will be evaluated using the grading system described by Fuchs-Buder. There are 4 items (jaw relaxation, vocal cord position, cough response, and limb movement) that are evaluated, and a total score can be calculated based on them: 1 point if all items are E, 3 points if even one item is P, and 2 points for the rest. A tracheal intubation condition rating of 1 or 2 indicates that the intubation is acceptable (successful), and a rating of 3 indicates that the intubation is unacceptable (unsuccessful).

SECONDARY OUTCOMES:
The rating of each item of the grading system of the tracheal intubation condition | During the tracheal intubation
  There are 4 items (jaw relaxation, vocal cord position, cough response, and limb movement) in the grading system described by Fuchs-Buder. We will also evaluate the grade of these items.
Total dose of remifentanil administered until tracheal intubation | From the start of the anesthesia induction to tracheal intubation
Incidence of hypotension and bradycardia | From the start of the anesthesia induction to tracheal intubation
Doses of agents (ephedrine and atropine) administered to treat hypotension and bradycardia | From the start of the anesthesia induction to tracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Sung Hye Byun, Daegu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng S, Xu Z, Wei Y, Zeng M, He J. Effect of intraoperative neuromonitoring on recurrent laryngeal nerve palsy rates after thyroid surgery--a meta-analysis. J Formos Med Assoc. 2013 Aug;112(8):463-72. doi: 10.1016/j.jfma.2012.03.003. Epub 2012 Sep 7. PMID 24016611
- [Background] Marusch F, Hussock J, Haring G, Hachenberg T, Gastinger I. Influence of muscle relaxation on neuromonitoring of the recurrent laryngeal nerve during thyroid surgery. Br J Anaesth. 2005 May;94(5):596-600. doi: 10.1093/bja/aei110. Epub 2005 Feb 25. PMID 15734779
- [Background] Combes X, Andriamifidy L, Dufresne E, Suen P, Sauvat S, Scherrer E, Feiss P, Marty J, Duvaldestin P. Comparison of two induction regimens using or not using muscle relaxant: impact on postoperative upper airway discomfort. Br J Anaesth. 2007 Aug;99(2):276-81. doi: 10.1093/bja/aem147. Epub 2007 Jun 15. PMID 17573390
- [Background] Lu IC, Wu SH, Wu CW. Neuromuscular blockade management for intraoperative neural monitoring. Kaohsiung J Med Sci. 2020 Apr;36(4):230-235. doi: 10.1002/kjm2.12153. Epub 2019 Nov 12. PMID 31713975
- [Background] Grant S, Noble S, Woods A, Murdoch J, Davidson A. Assessment of intubating conditions in adults after induction with propofol and varying doses of remifentanil. Br J Anaesth. 1998 Oct;81(4):540-3. doi: 10.1093/bja/81.4.540. PMID 9924229